CLINICAL TRIAL: NCT05661305
Title: Aswan Heart Centre - Egyptian Healthy Volunteers
Acronym: AHC-EHVol
Status: Recruiting | Type: Observational
Sponsor: Magdi Yacoub Heart Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AHC-EHVol
Record Dates: First submitted 2022-12-14; First posted 2022-12-22 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Genetic Predisposition to Disease
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood for whole genome sequencing.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Healthy Egyptian individuals to provide the first of its kind resource on human genetic variation in Egyptians, which is essential for understanding the significance of detected variations in patients with inherited cardiovascular disease and their families.
  Interventions: Other: Whole Genome Sequencing to compare healthy volunteers genome with that of cardiomyopathies patients.
- Cases: Egyptian patients and their family members diagnosed with different types hereditary cardiomyopathies.
  Interventions: Other: Whole Genome Sequencing to compare healthy volunteers genome with that of cardiomyopathies patients.

INTERVENTIONS:
Other: Whole Genome Sequencing to compare healthy volunteers genome with that of cardiomyopathies patients. — Egyptian patients and their family members diagnosed with different types hereditary cardiomyopathies.Healthy Egyptian individuals to provide the first of its kind resource on human genetic variation in Egyptians, which is essential for understanding the significance of detected variations in patients with inherited cardiovascular disease and their families.

SUMMARY:
To define the genotype of a healthy Egyptian cohort as a crucial step in determining the possible clinical implications of mutations detected in patients recruited in the registry.

DETAILED DESCRIPTION:
A key objective of the existing Cardiomyopathies project is to develop and validate assays to identify the genetic and molecular determinants of inherited cardiomyopathies in the Egyptian population.

Current sequencing technology has made cost- and time-effective whole exome and whole genome sequencing feasible. In their attempt to make clinically-relevant conclusions, genetecists, clinicians and bioinformaticians are increasingly faced by thousands of polymorphisms and variants, the clinical significance of which requires careful and systematic analysis of a number of factors including location of the mutation within the genome, type of mutation, gene affected and the protein for which it codes, functional importance of the coded protein, segregation within the family as well as frequency of the detected variation in the same population.

The latter step requires defining what constitutes the "genetic norm" (including normal variants) within the reference population. Data for different populations is already available in a number of databases that are accessible to the scientific community to help maximize the public benefit from research. Examples include the Exome Aggregation Consortium (ExAC) - which aggregates exome sequencing data from 60,706 unrelated individuals - and the 1000 Genomes Project which aggregates whole genome sequencing data from 2500 individuals.

However, to be able to confirm novel gene variants in the Egyptian population, data has to be compared to genomes of healthy individuals in the same population.

ELIGIBILITY:
* Inclusion Criteria:

  * Any adult Egyptian citizen subject that considers him/herself free of cardiovascular disease.
* Exclusion Criteria:

  * Individuals under 18 years of age
  * Known cardiovascular disease
  * Known collagen vascular disease
  * Individuals with communication difficulties, or who do not wish to participate
  * Pregnancy
  * Contraindication to MRI
  * Family history of sudden death
  * Family history of a familial cardiomyopathy
  * Family history of premature coronary artery disease (males <40 years, females <50 years).
* Withdrawal Criteria:

  * Withdrawal of consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1000 adult Egyptian citizen subjects that considers themselves free of cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Human genetic variation in Egyptians | 10 years
  To perform whole exome sequencing in 1000 healthy Egyptian individuals to provide the first of its kind resource on human genetic variation in Egyptians, which is essential for understanding the significance of detected variations in patients with inherited cardiovascular disease and their families.

CONTACTS AND LOCATIONS:
Overall Officials: Magdi H Yacoub, FRS OM, Principal Investigator — Imperial College London, and Magdi Yacoub Heart Foundation
Locations (1):
- Aswan Heart Centre - Magdi Yacoub Heart Foundation, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tan HL, Hofman N, van Langen IM, van der Wal AC, Wilde AA. Sudden unexplained death: heritability and diagnostic yield of cardiological and genetic examination in surviving relatives. Circulation. 2005 Jul 12;112(2):207-13. doi: 10.1161/CIRCULATIONAHA.104.522581. Epub 2005 Jul 5. PMID 15998675
- [Background] Lindgren A. Stroke genetics: a review and update. J Stroke. 2014 Sep;16(3):114-23. doi: 10.5853/jos.2014.16.3.114. Epub 2014 Sep 30. PMID 25328870
- [Background] UK10K Consortium; Walter K, Min JL, Huang J, Crooks L, Memari Y, McCarthy S, Perry JR, Xu C, Futema M, Lawson D, Iotchkova V, Schiffels S, Hendricks AE, Danecek P, Li R, Floyd J, Wain LV, Barroso I, Humphries SE, Hurles ME, Zeggini E, Barrett JC, Plagnol V, Richards JB, Greenwood CM, Timpson NJ, Durbin R, Soranzo N. The UK10K project identifies rare variants in health and disease. Nature. 2015 Oct 1;526(7571):82-90. doi: 10.1038/nature14962. Epub 2015 Sep 14. PMID 26367797
- [Background] 1000 Genomes Project Consortium; Auton A, Brooks LD, Durbin RM, Garrison EP, Kang HM, Korbel JO, Marchini JL, McCarthy S, McVean GA, Abecasis GR. A global reference for human genetic variation. Nature. 2015 Oct 1;526(7571):68-74. doi: 10.1038/nature15393. PMID 26432245
- [Background] Sudmant PH, Rausch T, Gardner EJ, Handsaker RE, Abyzov A, Huddleston J, Zhang Y, Ye K, Jun G, Fritz MH, Konkel MK, Malhotra A, Stutz AM, Shi X, Casale FP, Chen J, Hormozdiari F, Dayama G, Chen K, Malig M, Chaisson MJP, Walter K, Meiers S, Kashin S, Garrison E, Auton A, Lam HYK, Mu XJ, Alkan C, Antaki D, Bae T, Cerveira E, Chines P, Chong Z, Clarke L, Dal E, Ding L, Emery S, Fan X, Gujral M, Kahveci F, Kidd JM, Kong Y, Lameijer EW, McCarthy S, Flicek P, Gibbs RA, Marth G, Mason CE, Menelaou A, Muzny DM, Nelson BJ, Noor A, Parrish NF, Pendleton M, Quitadamo A, Raeder B, Schadt EE, Romanovitch M, Schlattl A, Sebra R, Shabalin AA, Untergasser A, Walker JA, Wang M, Yu F, Zhang C, Zhang J, Zheng-Bradley X, Zhou W, Zichner T, Sebat J, Batzer MA, McCarroll SA; 1000 Genomes Project Consortium; Mills RE, Gerstein MB, Bashir A, Stegle O, Devine SE, Lee C, Eichler EE, Korbel JO. An integrated map of structural variation in 2,504 human genomes. Nature. 2015 Oct 1;526(7571):75-81. doi: 10.1038/nature15394. PMID 26432246